CLINICAL TRIAL: NCT01779024
Title: Effects of Ghrelin on Alcohol Administration in Non-Treatment Seeking Heavy Drinkers
Brief Title: Ghrelin for Alcohol Use in Non-Treatment-Seeking Heavy Drinkers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 130043; 13-AA-0043
Record Dates: First submitted 2013-01-24; First posted 2013-01-29 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2017-06-01

CONDITIONS: fMRI; Alcohol Drinking; Alcoholism
Keywords: Addiction; Alcohol; Alcohol Clamp
MeSH Terms: conditions — Alcohol Drinking; Alcoholism; Behavior, Addictive | interventions — Ghrelin; Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ASA/Ghrelin (Experimental): Intravenous acyl-ghrelin [a loading dose (3 mcg/kg), followed by a continous infusion (16.9 ng/kg/min)] was administered on the first ASA visit; Intravenous placebo [packed in Dextrose 5% / Water USP 50mL bags and made identical to ghrelin in terms of appearance, texture, and odor] was administered on the second ASA visit.
  Interventions: Drug: Ghrelin; Drug: Alcohol
- ASA/Placebo (Placebo Comparator): Intravenous placebo [packed in Dextrose 5% / Water USP 50mL bags and made identical to ghrelin in terms of appearance, texture, and odor] was administered on the first ASA visit; Intravenous acyl-ghrelin [a loading dose (3 mcg/kg), followed by a continous infusion (16.9 ng/kg/min)] was administered on the second ASA visit
  Interventions: Drug: Placebo; Drug: Alcohol
- fMRI/Ghrelin (Experimental): Intravenous acyl-ghrelin [a loading dose (3 mcg/kg), followed by a continous infusion (16.9 ng/kg/min)] was administered on the first fMRI visit; Intravenous placebo [packed in Dextrose 5% / Water USP 50mL bags and made identical to ghrelin in terms of appearance, texture, and odor] was administered on the second fMRI visit.
  Interventions: Drug: Ghrelin; Procedure: fMRI
- fMRI/Placebo (Placebo Comparator): Intravenous placebo [packed in Dextrose 5% / Water USP 50mL bags and made identical to ghrelin in terms of appearance, texture, and odor] was administered on the first fMRI visit; Intravenous acyl-ghrelin [a loading dose (3 mcg/kg), followed by a continous infusion (16.9 ng/kg/min)] was administered on the second fMRI visit
  Interventions: Drug: Placebo; Procedure: fMRI

INTERVENTIONS:
Drug: Ghrelin
  Arms: ASA/Ghrelin; fMRI/Ghrelin
Drug: Placebo
  Arms: ASA/Placebo; fMRI/Placebo
Procedure: fMRI
  Arms: fMRI/Ghrelin; fMRI/Placebo
Drug: Alcohol
  Arms: ASA/Ghrelin; ASA/Placebo

SUMMARY:
Background:

- Ghrelin is a hormone in the human body that is mostly produced by the stomach. It makes people feel hungry, and also is connected with the desire to drink alcohol. Researchers want to test ghrelin to see if it can be used to control alcohol cravings and use. They will compare doses of ghrelin with a placebo in people who drink heavily.

Objectives:

- To study the effects of ghrelin on alcohol craving and use.

Eligibility:

* Individuals between 21 and 60 years of age who are heavy drinkers but are not seeking treatment for alcohol use.
* Participants must on average have more than 20 drinks per week for men, and more than 15 drinks per week for women.

Design:

* Participants will have a screening visit, four 2-night study visits, and a follow-up visit.
* Participants will be screened with a physical exam and medical history. They will provide urine and breath samples for drug testing. They will also answer questions about mood and physical symptoms, and about alcohol and other cravings.
* At the study visits, participants will stay overnight at the National Institutes of Health clinical center. They will spend the night at the center, have tests on the next day, and go home on the following morning. At each visit, participants will receive a ghrelin or placebo infusion, and will complete a series of tasks.
* For the first and second study visits, participants will have tests of alcohol craving and use. They will be able to receive alcohol infusions through a computer program that tests response time and craving reactions. At the same time, they will have a ghrelin or a placebo infusion. Blood alcohol levels, reaction time, and craving will be studied.
* For the third and fourth study visits, participants will have a magnetic resonance imaging (MRI) study. They will have an initial MRI to provide a picture of the brain. They will then have a functional MRI during which they will respond to a computer test. The test will allow them to win points for snack food or alcohol. This test will look at the brain s response time and craving reactions.
* There will be a follow-up visit 1 week after the fourth study visit. Some of the tests from the screening visit will be repeated.

DETAILED DESCRIPTION:
Objective:

Ghrelin is a 28-amino acid peptide acting as the endogenous ligand for the growth hormone secretagogue receptor (GHS-R). Ghrelin stimulates appetite by acting on the hypothalamic arcuate nucleus (ARC), a region that controls the intake of food and other substances, including alcohol. In addition to the ARC, GHS receptors (GHS-Rs) are also highly expressed in the caudal brain stem, the ventral tegmental area (VTA), hippocampus, substantia nigra, and dorsal and medial raphe nuclei. The expression of the GHS-R in the mesolimbic dopamine (DA) pathway suggests that ghrelin could play a role in reward processing. The role of ghrelin in the DA reward processing and the role of the DA reward system in alcoholism suggest a role of ghrelin in alcoholism. Consistent with this hypothesis, preclinical studies demonstrate that both ghrelin and ethanol activate the cholinergic-dopaminergic reward link, implying neurochemical analogies between ghrelin and ethanol. This supports the hypothesis that ghrelin is involved in mediating the rewarding properties of ethanol. Additional animal experiments demonstrate that the central ghrelin action not only stimulates the reward processing but is also required for stimulation of that system by alcohol. Human studies show reduced ghrelin levels in actively drinking alcoholics; increased ghrelin levels during alcohol abstinence; and a positive correlation between ghrelin level and alcohol craving scores. More recently, a study conducted at Brown University by the PI demonstrated the safety of the administration IV of human ghrelin to non-treatment seeking alcohol-dependent heavy drinking individuals. Furthermore, a preliminary interim analysis shows that IV ghrelin administration may lead to a temporary significant increase in alcohol craving. The primary objective of this protocol is to investigate whether IV ghrelin, as compared to placebo, will increase motivation for alcohol reward, as measured by a progressive ratio (PR) schedule paradigm with IV alcohol self-infusion (primary aim). We will also assess a number of secondary aims. Specifically, we will also assess whether IV ghrelin, as compared to placebo, will also alter urges to drink and the subjective response to IV alcohol. Adverse events will also be assessed to ensure the safety of the IV coadministration of ghrelin and alcohol. During an fMRI/alcohol clamp session, fMRI will be used to see whether ghrelin affects the activation of the ventral striatum induced by acute IV alcohol administration and the incentive salience of cues associated with alcohol administration.

Study Population:

Male and female participants will be non-treatment seeking heavy drinking volunteers.

Design:

The study is designed as a within-subject, double-blind, placebo-controlled study of ghrelin. The first visit will be the initial screening visit. The second and third visits will be PR sessions with IV ethanol, during which each participant will also receive IV ghrelin (or matched placebo). The fourth and fifth visits will combine an fMRI session with an alcohol clamp session (i.e. a fixed dose of alcohol will be administered) and subjects will participate in a modified version of the monetary incentive delay (MID) task in which they will respond to cues that indicate the opportunity to press a button to gain a reward. On some trials the reward will be points that can be exchanged for snack foods while on other trials the reward will be points that will determine how much intravenous alcohol a subject will be given during the alcohol clamp procedure which will immediately follow the modified MID task. After the modified MID task is complete subjects will have a short break and then begin the alcohol IV infusion.

Outcome measures:

The primary measure of this study will be the breakpoint, which is the schedule (number of button presses) at which the individual stops to work for more alcohol. Also, the BrAC exposure measures will be determined. Alcohol craving in response to ghrelin will be measured using the Alcohol Visual Analogue Scale (A-VAS) and the Alcohol Urge Questionnaire (AUQ) during the PR sessions. Sensitivity to alcohol will be measured using the Drug Effects Questionnaire (DEQ), Biphasic Alcohol Effects Scale (BAES), and the Profile of Mood States (POMS), repeatedly during the PR sessions and the CASE Experience Questionnaire (CEQ) at the end of all sessions. fMRI BOLD signal in brain areas associated with incentive salience and areas associated with reward circuitry (including the ventral striatum) will be measured during the fMRI/alcohol clamp session. This study may facilitate the identification of a novel neuropharmacological target, thus facilitating the development of novel pharmacological treatments for alcoholism.

ELIGIBILITY:
* INCLUSION CRITERIA:

Male and female participants between 21-60 years of age.

Good health as determined by medical history, physical exam, ECG and lab tests.

Creatinine less than to 2 mg/dl.

Female must have a negative urine pregnancy (hCG) test at the start of each study session. Females of childbearing potential who are sexually active and have not been surgically sterilized must agree to use an adequate method of birth control during the study. Adequate methods of contraception for sexually active women are having a male sexual partner(s) who is surgically sterilized prior to inclusion; having a sexual partner(s) who is/are exclusively female; using oral contraceptives (either combined or progestrogen only) with a single-barrier method of contraception consisting of spermicide and condom or diaphragm; using double-barrier contraception, specifically, a condom plus spermicide and a female diaphragm or cervical cap plus spermicide; or using an approved intrauterine device (IUD) with established efficacy.

Participants must drink alcohol regularly at a heavy level, on average greater than 20 drinks per week for men, and greater than 15 drinks per week for women, and not be seeking help for alcohol-related problems.

Participant must be willing to receive two IV lines.

EXCLUSION CRITERIA:

Current or prior history of any clinically significant disease, including CNS, cardiovascular, respiratory, gastrointestinal, hepatic, renal, endocrine, or reproductive disorders.

Specific exclusion criteria related to the administration of ghrelin, are chronic inflammatory diseases (e.g., Crohn s disease, ulcerative colitis, celiac disease) diabetes, obesity (BMI greater than or equal 30 kg/m(2), weight greater than or equal to 120 Kg, high triglycerides level (> 350 mg/dL), history of clinically significant hypotension (e.g.: history of fainting and/or syncopal attacks) and/or resting systolic BP < 100 mmHg.

Positive hepatitis or HIV test at screening.

Current clinically significant major depression or anxiety; or prior clinically significant psychiatric problems, including eating disorders, schizophrenia, bipolar disorder, obsessive compulsive disorder.

Current diagnosis of substance dependence (other than alcohol or nicotine).

Currently seeking treatment for alcohol use disorder.

History of significant withdrawal symptoms or presence of clinically significant withdrawal symptoms (Clinical Institute Withdrawal Assessment (CIWA) score > 8) at screening.

Non-drinkers (alcohol-naive individuals or current abstainers) or no experience drinking 5 or more drinks on one occasion.

Unable to provide a negative urine drug screen.

Pregnancy or intention to become pregnant for women. Female participants will undergo a urine beta-hCG test to ensure they are not pregnant.

Use of prescription or OTC medications known to interact with alcohol within 2 weeks of the study. These include, but may not be limited to: isosorbide, nitroglycerine, benzodiazepines, warfarin, anti-depressants such as amitriptyline, clomipramine and nefazodone, anti-diabetes medications such as glyburide, metformin and tolbutamide, H2-antagonists for heartburn such as cimetidine and ranitidine, muscle relaxants, anti-epileptics including phenytoin and Phenobarbital codeine, and narcotics including darvocet, percocet and hydrocodone. Drugs known to inhibit or induce enzymes that metabolize alcohol should not be used for 4 weeks prior to the study. These include chlorzoxazone, isoniazid, metronidazole and disulfiram. Cough-and-cold preparations, which contain antihistamines, pain medicines and anti-inflammatories such as aspirin, ibuprofen, acetaminophen, celecoxib and naproxen, should be withheld for at least 72 hours prior to each study session.

Current or prior history of alcohol-induced flushing reactions.

Contraindications for MRI scanning, including metal in body that are contraindicated for MRI (such as implants, pacemaker, prostheses, shrapnel, irremovable piercings), left-handedness, and claustrophobia.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2012-12-13; Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Leggio, M.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kojima M, Hosoda H, Date Y, Nakazato M, Matsuo H, Kangawa K. Ghrelin is a growth-hormone-releasing acylated peptide from stomach. Nature. 1999 Dec 9;402(6762):656-60. doi: 10.1038/45230. PMID 10604470
- [Background] Cummings DE, Naleid AM, Figlewicz Lattemann DP. Ghrelin: a link between energy homeostasis and drug abuse? Addict Biol. 2007 Mar;12(1):1-5. doi: 10.1111/j.1369-1600.2007.00053.x. No abstract available. PMID 17407491
- [Background] Jerlhag E, Egecioglu E, Dickson SL, Andersson M, Svensson L, Engel JA. Ghrelin stimulates locomotor activity and accumbal dopamine-overflow via central cholinergic systems in mice: implications for its involvement in brain reward. Addict Biol. 2006 Mar;11(1):45-54. doi: 10.1111/j.1369-1600.2006.00002.x. PMID 16759336
- [Background] Leggio L, Zywiak WH, Fricchione SR, Edwards SM, de la Monte SM, Swift RM, Kenna GA. Intravenous ghrelin administration increases alcohol craving in alcohol-dependent heavy drinkers: a preliminary investigation. Biol Psychiatry. 2014 Nov 1;76(9):734-41. doi: 10.1016/j.biopsych.2014.03.019. Epub 2014 Mar 25. PMID 24775991
- [Background] Leggio L, Schwandt ML, Oot EN, Dias AA, Ramchandani VA. Fasting-induced increase in plasma ghrelin is blunted by intravenous alcohol administration: a within-subject placebo-controlled study. Psychoneuroendocrinology. 2013 Dec;38(12):3085-91. doi: 10.1016/j.psyneuen.2013.09.005. Epub 2013 Sep 13. PMID 24090583
- [Background] Leggio L, Ferrulli A, Cardone S, Nesci A, Miceli A, Malandrino N, Capristo E, Canestrelli B, Monteleone P, Kenna GA, Swift RM, Addolorato G. Ghrelin system in alcohol-dependent subjects: role of plasma ghrelin levels in alcohol drinking and craving. Addict Biol. 2012 Mar;17(2):452-64. doi: 10.1111/j.1369-1600.2010.00308.x. Epub 2011 Mar 11. PMID 21392177
- [Background] Leggio L. Role of the ghrelin system in alcoholism: Acting on the growth hormone secretagogue receptor to treat alcohol-related diseases. Drug News Perspect. 2010 Apr;23(3):157-66. doi: 10.1358/dnp.2010.23.3.1429490. PMID 20440417
- [Result] Farokhnia M, Grodin EN, Lee MR, Oot EN, Blackburn AN, Stangl BL, Schwandt ML, Farinelli LA, Momenan R, Ramchandani VA, Leggio L. Exogenous ghrelin administration increases alcohol self-administration and modulates brain functional activity in heavy-drinking alcohol-dependent individuals. Mol Psychiatry. 2018 Oct;23(10):2029-2038. doi: 10.1038/mp.2017.226. Epub 2017 Nov 14. PMID 29133954
- [Derived] Richardson RS, Farokhnia M, Vendruscolo LF, Leggio L. Plasma concentrations of the inflammatory adipokine lipocalin-2 are not affected by chronic alcohol exposure in rats or acute alcohol administration in people with alcohol use disorder. Am J Drug Alcohol Abuse. 2025;51(6):730-740. doi: 10.1080/00952990.2025.2582563. Epub 2025 Dec 2. PMID 41329966

RESULTS

PARTICIPANT FLOW:
Groups:
- Ghrelin, Then Placebo: Intravenous acyl-ghrelin a loading dose (3 mcg/kg), followed by a continuous infusion (16.9 ng/kg/min)] was administered on the first visit; Intravenous placebo [packed in Dextrose 5% / Water USP 50mL bags and made identical to ghrelin in terms of appearance, texture, and odor] was administered on the second visit.
- Placebo, Then Ghrelin: Intravenous placebo packed in Dextrose 5% / Water USP 50mL bags and made identical to ghrelin in terms of appearance, texture, and odor] was administered on the first visit; Intravenous acyl-ghrelin [a loading dose (3 mcg/kg), followed by a continuous infusion (16.9 ng/kg/min)] was administered on the second visit
Period: 1st Visit - Alcohol Self-Administration
Arm/Group | Ghrelin, Then Placebo | Placebo, Then Ghrelin
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0
Period: 2nd Visit - Alcohol Self-Administration
Arm/Group | Ghrelin, Then Placebo | Placebo, Then Ghrelin
Started | 8 | 9
Completed | 6 | 9
Not Completed | 2 | 0
Period: 1st Visit - Functional MRI
Arm/Group | Ghrelin, Then Placebo | Placebo, Then Ghrelin
Started | 6 | 7
Completed | 4 | 5
Not Completed | 2 | 2
Period: 2nd Visit - Functional MRI
Arm/Group | Ghrelin, Then Placebo | Placebo, Then Ghrelin
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either Ghrelin or Placebo
Arm/Group | All Study Participants
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 2
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Infusions Self-administered
Description: The total number of alcohol infusions self-administered.
Time Frame: 120 minutes after the start of the infusion
Population: The analyses included only those subjects who completed all types of infusions (Ghrelin and Placebo) and had alcohol self-administration
Measure: Mean (Standard Error); unit: Number of alcohol infusions
Groups:
- Ghrelin: Intravenous acyl-ghrelin a loading dose (3 mcg/kg), followed by a continous infusion (16.9 ng/kg/min)] was administered on the first ASA visit; Intravenous placebo [packed in Dextrose 5% / Water USP 50mL bags and made identical to ghrelin in terms of appearance, texture, and odor] was administered on the second ASA visit.
- Placebo: Intravenous placebo packed in Dextrose 5% / Water USP 50mL bags and made identical to ghrelin in terms of appearance, texture, and odor] was administered on the first ASA visit; Intravenous acyl-ghrelin [a loading dose (3 mcg/kg), followed by a continous infusion (16.9 ng/kg/min)] was administered on the second ASA visit
Arm/Group | Ghrelin | Placebo
Number analyzed (Participants) | 11 | 11
Number of alcohol infusions | 10.45 (1.15) | 8.80 (1.29)

ADVERSE EVENTS:
Time Frame: 240 minutes
Groups:
- Ghrelin: Intravenous acyl-ghrelin a loading dose (3 mcg/kg), followed by a continous infusion (16.9 ng/kg/min)] was administered on the first visit; Intravenous placebo [packed in Dextrose 5% / Water USP 50mL bags and made identical to ghrelin in terms of appearance, texture, and odor] was administered on the second visit.
- Placebo: Intravenous placebo packed in Dextrose 5% / Water USP 50mL bags and made identical to ghrelin in terms of appearance, texture, and odor] was administered on the first visit; Intravenous acyl-ghrelin [a loading dose (3 mcg/kg), followed by a continous infusion (16.9 ng/kg/min)] was administered on the second visit
Arm/Group | Ghrelin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 12/17 | 7/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ghrelin (N=17) | Placebo (N=17)
Dizziness (Cardiac disorders) | 2 | 4
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 0 | 1
Decreased appetite (General disorders) | 1 | 0
Fatigue (General disorders) | 5 | 1
Feeling hot (General disorders) | 1 | 0
Flushing (General disorders) | 1 | 0
Hyperhidrosis (General disorders) | 2 | 2
Increased Appetite (General disorders) | 10 | 5
Headache (Nervous system disorders) | 1 | 1
Memory impairment (Nervous system disorders) | 2 | 1
Somnolence (Nervous system disorders) | 7 | 6
Euphoric mood (Psychiatric disorders) | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT01779024/Prot_SAP_000.pdf